CLINICAL TRIAL: NCT02763085
Title: Clinical Evaluation of "Basic Filling" Material in Class I and II Cavities: A Prospective Controlled Clinical Trial up to 3 Years
Brief Title: Clinical Evaluation of Basic Filling Material in Class I and II Posterior Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Principal Investigator, Funda Ozturk Bozkurt, Dr., Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 283 (108400987-308)
Record Dates: First submitted 2016-02-14; First posted 2016-05-05 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Caries; Unsatisfactory Restoration of Tooth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Basic Filling Material (Experimental): Fillings made with a new dental filling material.
  Interventions: Device: Basic Filling Material

INTERVENTIONS:
Device: Basic Filling Material — Tooth (teeth) affected by dental caries or with an existing defective filling will be restored using the materials listed (Basic Filling Material). Procedures will be done using local anesthesia. The cavity is excavated and filled according to the guidelines for ordinary restorative techniques.
  Other Names: Dental Filling

SUMMARY:
Evaluation of a new basic filling restorative material.

In contemporary dentistry, clinicians have essentially three types of material choices for direct restorations: amalgam, resin composite, and glass ionomer restoratives.

Due to the toxicity of mercury and the subsequent environmental problems, the search for alternatives continues and search into new composite restorative materials intensifies. Recognized disadvantages of tooth colored resin based restorative materials are as polymerization shrinkage, postoperative sensitivity and technical procedure complexity. Higher rates of occlusal wear and lower toughness are disadvantages of glass ionomer restoratives.

Therefore, alternative materials are being developed to compensate the disadvantages of current contemporary tooth coloured restorative materials. Nevertheless, the search for simplification for restoring missing dental tissues introduced the "basic filling concept".

This project aims to study the clinical performance of this new basic filling restorative material for Class I and Class II cavities. 80 patients are recruited to the project which is carried out at the School of dentistry, Istanbul Medipol University, Turkey.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the clinical performance of a new basic filling restorative material for Class I and Class II cavities that needs to be restored in permanent teeth.

Basic filling material combines the handling properties of glass ionomer restorative materials with the mechanical properties of resin composite restorative materials.

Extensive laboratory studies have been performed on the new material, but the clinical attributes have yet to be disclosed.

The study will be carried out as a prospective study, with assessment of the restorations after three year.

The project includes 80 patients. Most of the patients have been recruited from the Istanbul Medipol University Dental Clinics in Istanbul.

After giving their consent to take part in the study Class I & II restorations of both upper and lower molars and premolars are performed

The treatment procedure is:

The patients are offered local anesthetic before treatment start. The cavity is excavated and filled according to the guidelines for composite restorations.

The control procedure is:

The restoration is evaluated according to marginal adaptation, cavo surface marginal discoloration, approximal contact, fractures, caries associated with restorations and postoperative hypersensitivity. The controls will take place after two weeks, one year, two years and three years.

ELIGIBILITY:
Inclusion Criteria:

* Vital tooth
* Caries removal or restoration replacement (i.e. amalgam, composite, glass-ionomer)
* Class I & II restorations premolar and molars
* Maximum 2 fillings with the Basic Filling material in each patient
* No obvious untreated caries, dental health problems (regularly checked by a dentist)
* Good or moderate oral hygiene (plaque score of less than 30% in anterior region before treatment)
* No untreated periodontal disease (only DPSI 1, 2)
* Subjects had to be over the age of 18, be classified according to the American Society of Anesthesiologists (ASA) as ASA I or ASA II, present with moderate to good oral hygiene, and be free of periodontal disease (probing depth and attachment levels within normal limits, no furcation involvement, and no mobility)

Exclusion Criteria:

* Caries extends cemento-enamel junction in Class II
* Considerable horizontal and/or vertical mobility of teeth: tooth mobility index score 2 or 3
* Considerable periodontal disease without treatment (DPSI 3-, 3+ and 4)
* Endodontic treatment
* Patients who still want to bleach their teeth or bleached teeth less than 3 weeks ago
* Excluding the teeth, without opposing natural dentition (either intact or restored with intracoronal or extracoronal fixed restorations), and with a minimum of 20 teeth
* Subjects who presented with severe wear facets and/or reported parafunctional activities such as clenching or nocturnal bruxism
* Subjects who were pregnant or breast feeding during the duration of the study
* Subjects who are known to be allergic to the ingredients of resin materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2018-09 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
FDI (World Dental Federation) criteria for dental restorations assessment | at 3 years
  2 independent evaluators The primary outcome will consist in the FDI (World Dental Federation) instrument for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010 . This instrument is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually.The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome.
  Hickel R, Peschke A, Tyas M, Mjör I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66.

SECONDARY OUTCOMES:
Plaque accumulation according to the Silness & Löe (1964) Plaque Index | at 3 years
  0 = No plaque in the gingival area.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent
Gingival Inflammation according to the Silness & Löe (1964) Gingival Index. | at 3 years
  0 = Normal gingival.
  1. = Mild inflammation-slight change in colour, slight oedema. No bleeding on probing
  2. = Moderate inflammation-redness, oedema and glazing. Bleeding on probing.
  3. = Severe inflammation-marked redness and oedema. Ulceration. Tendency to spontaneous bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Emir Yuzbasioglu, DDS,PhD, Principal Investigator — Medipol University; Mutlu Ozcan, DDS,PhD, Principal Investigator — University of Zurich
Locations (1):
- Istanbul Medipol University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No